CLINICAL TRIAL: NCT06665113
Title: A Double-blinded, Randomized, Parallel-group, Superiority Study to Explore the Neuroprotective Effects of Long-term Transcutaneous Auricular Vagus Nerve Stimulation(taVNS) in Early Parkinson's Disease(PD) Patients
Brief Title: Neuroprotective Effects of Long-term TaVNS in Early Parkinson's Disease Patients
Acronym: NLTVNSPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kezhong Zhang (Other)
Responsible Party: Sponsor-Investigator, Kezhong Zhang, Professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-SR-1019
Record Dates: First submitted 2024-10-20; First posted 2024-10-30 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Parkinson Disease, Idiopathic; Vagus Nerve Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard anti-Parkinson's disease medication treatment + taVNS real stimulation (Experimental): For the real stimulation group, two modified point electrodes will deliver stimulation near the auricular branch of the vagus nerve in the left concha cymba.
  Each Parkinson's disease patient will receive one 30-minute stimulation session per day(at least 5 days per week) for 270 consecutive days.
  Interventions: Device: taVNS real stimulation
- Standard anti-Parkinson's disease medication treatment + taVNS sham stimulation (Sham Comparator): For the sham stimulation group, two modified point electrodes will deliver stimulation to the earlobes.Each Parkinson's disease patient will receive one 30-minute stimulation session per day(at least 5 days per week) for 270 consecutive days.
  Interventions: Device: taVNS sham stimulation

INTERVENTIONS:
Device: taVNS real stimulation — For the real stimulation group, two modified point electrodes will deliver stimulation near the auricular branch of the vagus nerve in the left concha cymba. Stimulation parameters: frequency = 20 Hz; pulse width = 500 μs; continuous stimulation for 60 seconds, followed by a 10-second off period, repeated for 30 minutes.
  Arms: Standard anti-Parkinson's disease medication treatment + taVNS real stimulation
Device: taVNS sham stimulation — For the sham stimulation group, two modified point electrodes will deliver stimulation to the earlobes.Stimulation parameters: frequency = 20 Hz; pulse width = 500 μs; continuous stimulation for 60 seconds, followed by a 10-second off period, repeated for 30 minutes.
  Arms: Standard anti-Parkinson's disease medication treatment + taVNS sham stimulation

SUMMARY:
This study is a randomized, double-blind, controlled trial exploring the effects of long-term taVNS intervention in patients with early-stage Parkinson's disease.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, controlled trial exploring the effects of long-term taVNS intervention in patients with early-stage Parkinson's disease, , aiming to investigate a novel therapeutic approach for delaying PD progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-75 years.
2. Clinically diagnosed Idiopathic Parkinson's disease patients according to the 2016 Chinese diagnostic criteria for Parkinson's disease.
3. Hoehn and Yahr (H&Y) stage ≤ 2.5 at medication initiation.
4. Parkinson's disease duration ≤ 3 years.
5. Receiving standard anti-Parkinson's disease medication treatment.

Exclusion Criteria:

1. Patients with cognitive impairment (MMSE < 24 and/or MoCA < 26) or mental illnesses, or those unable to cooperate for other reasons.
2. Use of neuroprotective medications within 90 days prior to baseline, including monoamine oxidase B inhibitors (rasagiline, selegiline), certain dopamine receptor agonists (ropinirole), and GLP-1 receptor agonists such as Exenatide and NLY-01.
3. Use of any medications that may affect dopamine metabolism and/or dopamine receptors within 90 days prior to baseline, including typical and atypical antipsychotics, metoclopramide, α-methyl-dopa, flunarizine, apomorphine, amphetamine derivatives, bupropion, buprenorphine, cocaine, meperidine, methamphetamine, norephedrine, phentermine, modafinil, methylphenidate, procyclidine, reserpine, phenylpropanolamine, or MAO-A inhibitors.
4. Previous treatment with vagus nerve stimulation.
5. MRI contraindications (e.g., claustrophobia unresponsive to comfort or low-dose anxiolytics, dental implants) or MRI scans indicating clinically significant abnormalities in the brain, including but not limited to past hemorrhages or infarcts > 1 cm³ or > 3 lacunar infarcts.
6. Contraindications for taVNS, such as patients with cardiac pacemakers or a history of DBS surgery, or those planning surgery during the trial; ear conditions, such as tympanic membrane perforation.
7. Atypical or secondary Parkinsonian syndromes, including but not limited to those caused by trauma, brain tumors, infections, cerebrovascular diseases, or other neurological disorders, or symptoms confirmed by the investigator as drug, chemical, or toxin-related.
8. Previous history of stroke or intracranial mass lesions.
9. Patients with existing or potential cardiovascular diseases.
10. Ophthalmic diseases affecting eye movements.
11. Any neurological disorders other than Parkinsonian motor symptoms that interfere with gait or balance (e.g., chronic pain) or musculoskeletal injuries (e.g., fractures, stroke sequelae).
12. Severe organic diseases, such as late-stage tumors, with a life expectancy of less than 2 years.
13. Concurrent participation in other clinical trials.
14. Inability to receive the required treatment and follow-up due to geographic reasons.
15. Any subject with an upper limb UPDRS tremor score of 3 or higher.
16. Patients with a history of PD-related freezing episodes or falls.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
MDS-UPDRS-Ⅲ | baseline, 180±7 days, 360±7 days, 540±7 days，570±7 days
  Used to evaluate the motor function.
Free water in the posterior substantia nigra (DTI) | baseline, 180±7 days, 360±7 days, 540±7 days，570±7 days
  Used to measure progression of early Parkinson's disease.

SECONDARY OUTCOMES:
Scales: MDS-UPDRS-II | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Used to evaluate quality of life of PD.
Step Length、Stride Length、Stride Velocity and Step Length Variability | baseline,180±7 days, 360±7 days, 540±7 days，570±7 days
  Used to assess the patient's gait disturbances，including the Step Length、Stride Length、Stride Velocity and Step Length Variability
Scales: H&Y stage | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Used to evaluate the stage of PD.

OTHER OUTCOMES:
Eye-Tracking Technology | baseline,180±7 days, 360±7 days, 540±7 days，570±7 days
  Fixation Duration: The length of time the gaze remains on a single point. Saccade Velocity: The speed of eye movements between fixations. Scan Path: The trajectory of eye movements during visual exploration
Electroencephalogram (EEG) | baseline,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Brain wave activity (measured in microvolts, µV).
MRI | baseline,180±7 days, 360±7 days, 540±7 days，570±7 days
  T1-weighted Imaging:
  Measurement: Structural brain volume (measured in cubic centimeters, cm³).
  BOLD fMRI:
  Measurement: Blood oxygen level-dependent signals (measured in percentage change).
  Diffusion Tensor Imaging (DTI):
  Fractional Anisotropy (FA):
  Measurement: FA values (unitless, scale from 0 to 1).
  Mean Diffusivity (MD):
  Measurement: MD values (measured in mm²/s).
  NM-MRI:
  Measurement: Neurochemical markers (unit as appropriate).
  Iron-sensitive MRI:
  Quantitative Susceptibility Mapping (QSM):
  Measurement: Susceptibility values (measured in parts per million, ppm).
  Susceptibility Weighted Imaging (SWI):
  Measurement: Signal intensity (unitless).
  R2*:
  Measurement: Relaxation rate (measured in Hz).
Number of participants with the following Serum biomarkers: | baseline,180±7 days, 360±7 days, 540±7 days，570±7 days
  Brain-Derived Neurotrophic Factor (BDNF):
  Measurement: Concentration (measured in ng/mL).
  Glial Fibrillary Acidic Protein (GFAP):
  Measurement: Concentration (measured in ng/mL).
  Neurofilament Light Chain (NFL):
  Measurement: Concentration (measured in pg/mL).
  Tau Protein:
  Measurement: Concentration (measured in pg/mL).
  Tumor Necrosis Factor Alpha (TNF-α):
  Measurement: Concentration (measured in pg/mL).
  Interleukin-6 (IL-6):
  Measurement: Concentration (measured in pg/mL).
  Interleukin-1 Beta (IL-1β):
  Measurement: Concentration (measured in pg/mL).
Movement Disorder Society Unified Parkinson's Disease Rating Scale - Part I (MDS-UPDRS-I) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  .Measurement: Score (range: 0-52; higher score indicates worse non-motor function).
Non-Motor Symptoms Scale (NMSS) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-100; higher score indicates more severe non-motor symptoms).
Activities of Daily Living (ADL) Scale | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-100; higher score indicates greater independence).
Hamilton Anxiety Scale (HAMA) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-56; higher score indicates greater anxiety).
Hamilton Depression Rating Scale - 24 items (HAMD-24) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-76; higher score indicates greater depression severity).
Apathy Scale (AS) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-42; higher score indicates greater apathy).
Rapid Eye Movement Sleep Behavior Disorder Questionnaire (RBDSQ) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-25; higher score indicates more severe symptoms).
Epworth Sleepiness Scale (ESS) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-24; higher score indicates greater daytime sleepiness).
Montreal Cognitive Assessment (MoCA) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-30; higher score indicates better cognitive function).
Hopkins Verbal Learning Test - Revised (HVLT-R) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (varies by subscale; higher score indicates better verbal memory).
Judgment of Line Orientation (JLO) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-30; higher score indicates better visual-spatial abilities).
Letter-Number Sequencing (LNS) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (range: 0-30; higher score indicates better working memory).
Symbol Digit Modalities Test (SDMT) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Score (varies based on response time; higher score indicates faster processing speed).
Levodopa Equivalent Dose (LED) | baseline,30±3 days,90±5 days,180±7 days, 360±7 days, 540±7 days，570±7 days
  Measurement: Dose (measured in mg; higher dose indicates greater medication requirement).

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, Professor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No